CLINICAL TRIAL: NCT02176785
Title: The Effect of Pre-Frontal tDCS on Sleep Propensity During an Afternoon Nap: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Power Nap
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-05

CONDITIONS: Sleep
Keywords: Sleep; Transcranial Electric Stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham tDCS (Sham Comparator): tDCS will be applied, but then turned off after 30 seconds.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- Anodal tDCS 2mA 10 Minutes (Experimental): Anodal tDCS will be applied bi-frontally for 10 minutes at 2mA
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- Cathodal tDCS 2mA 10 Minutes (Experimental): Cathodal tDCS will be applied Bi-Frontally for 10 minutes at 2mA
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — tDCS will be delivered using a Chattanooga Ionto™ Iontophoresis System - Phoresor.
  Other Names: Chattanooga Ionto™ Iontophoresis System - Phoresor.

SUMMARY:
Transcranial Direct Current Stimulation (tDCS) is a safe, non-invasive brain stimulation technology that has demonstrated the ability to temporarily increase or decrease activity in specific regions of the brain. The researchers are investigating the effect of this technology on sleep propensity by applying two different types of stimulation as well as sham (Placebo) stimulation during three different afternoon naps. The researchers are subsequently hoping to recruit healthy volunteers without medical, or sleep problems who have a regular sleep schedule to participate in the study

DETAILED DESCRIPTION:
Recent studies have demonstrated that there are cortical direct current (DC) changes that accompany sleep onset and transitions between sleep states in a stereotyped manner. In these studies it was determined that negative potential shifts occurred prior to and at the transition from wakefulness to sleep and at transitions between Rapid Eye Movement sleep (REM) sleep, and Non-Rapid Eye Movement (NREM) sleep. In a subset of experiments it was demonstrated that the same DC potential shifts occur during the transition from wake to sleep in an afternoon nap. The recorded DC potential shifts occurred predominantly in the pre-frontal cortex (F3, F4), with spread into central areas. No current literature exists that explores whether tDCS could be used to modulate cortical activity prior to sleep, resulting in either increased or decreased sleep propensity.

The application of focal, non-invasive brain stimulation has already led to novel and effective treatments for neuropsychiatric disease with minimal side effects (Most well studied in depression and repetitive Transcranial Magnetic Stimulation or, rTMS). Should the application of tDCS modulate sleep propensity it would represent a novel study paradigm with the potential to lead to a completely novel treatment for sleep disturbance. With this small pilot study, we propose taking the first step in exploring the utility of tDCS in modulating sleep propensity. We propose to recruit 15 healthy non-treatment seeking participants from the community and expose them to three total nap conditions in a randomized counter balanced fashion, with 10 minutes of either, Anodal, Cathodal, or Sham tDCS stimulation occurring prior to each nap opportunity.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* capable of coming in for an initial intake screen, and then again for 2 hours on consecutive Monday, Wednesday, and Friday afternoons

Exclusion Criteria:

* Presence of Neurologic, psychiatric, or sleep disorder.
* Current use of medications affecting the central nervous system.
* Daily consumption of alcohol, or consequences of alcohol use (DUI, occupational, or social dysfunction ect.).
* Tobacco use.
* Consumption of more than the equivalent of 300mg of caffeine daily.
* Habitual sleep duration of less than 6 ½ hours, greater than 8 ½ hours, a difference between weeknight, and weekend sleep of greater than 3 hours, or typical sleep timing more than 3 hours outside of the window of 10pm-6am.
* Score of greater than 5 on the Pittsburgh Sleep Quality Index (PSQ-I), or 10 on the Epworth Sleepiness scale (ESS).
* BMI greater than 30, or Heavy snoring.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sleep onset latency and sleep architecture | 30 Minutes
  Sleep onset latency and sleep architecture will be assessed using polysomnography during a 30 minute nap opportunity.

SECONDARY OUTCOMES:
Sleep quality | 30 Minutes
  Sleep quality will be assessed with a visual analog scale following each nap opportunity.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States